CLINICAL TRIAL: NCT01775956
Title: A Retrospective Review of a Comprehensive Cohort of Septic Shock: Assessment of Critical Determinants of Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Anand Kumar, MD, University of Manitoba
Other Study IDs: H2003:087
Record Dates: First submitted 2013-01-16; First posted 2013-01-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Septic shock remains the dominant cause of death in ICU's of the developed world with approximately 400,000 cases annually in the US and another 20,000 annually in Canada. While many retrospective and prospective reviews of septic shock patients have been undertaken worldwide, many key questions remain unanswered. These questions include the true incidence, associated morbidity and mortality of septic shock in North America, key factors associated with successful management and markers suggesting a high probability of a complicated clinical course. Part of the reason for the persistence of these questions, is the fact that previous and ongoing reviews of septic shock and severe sepsis have been either limited in number (typically <150) or biased by the need to be eligible for specific clinical trials (typically, non-eligible patients have not been followed and had data collected.

We propose to examine specific questions within a temporally comprehensive cohort of septic shock patients by review of individual charts using a defined data-extraction template.

DETAILED DESCRIPTION:
Objectives

* Determination of impact of rapidity of implementation of antibiotic therapy, source control (where required) and fluid resuscitation on mortality of septic shock
* Utility of persistence or increase of vasopressor needs over the 1st 24 hours of shock as a predictor of a complicated ICU course (ICU duration > 1 week) or death
* Assessment of initial biochemical parameters, co-morbidities and new onset organ failure at admission as predictors of a complicated ICU course (ICU duration > 1 week) and death

Data Collection: Data collection would be performed by a combination of study nurses and 2nd or 3rd year medical students hired for the summer for this research project. Research nurses and student will be trained by the principal investigator. A minimum of 10% of the charts will be randomly audited by the principal investigator to ensure appropriate data extraction. This will allow the PI to review and correct any discrepant coding issues and judge specific questions (e.g. appropriateness of antibiotics/presence of effective antibiotics or not).

Data Collection Tool: Attached. In addition, data in the ICU registry includes basic epidemiologic data (age, sex, all pertinent medical/surgical comorbidities/risk factors, etc) as well as all Apache II

ELIGIBILITY:
Inclusion criteria.

* The primary analysis will include all patients admitted to the institution with a final diagnosis of septic shock (including transfers).

Exclusion criteria:

* ICU patients who do not have a diagnosis of septic shock
* These are the only Inclusion/Exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical charts from all patients coded as septic shock in an internal ICU registry since 1994.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2003-12; Primary Completion 2018-01 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Outcome as determined by treatment choices | Participants will be followed for the Average length of hospital stay 4-5 weeks
  Analysis will be used to examine critical therapeutic elements of outcome (choice of antibiotics, rapidity of initiation, use of multiple drug combinations, choice and speed of initiation of pressors, choice and degree of fluid resuscitation, etc).
  Preliminary analysis of data from 2800 charts suggests an annual incidence of incidence of septic shock in North America (without adjustment for age, sex or socioeconomic status) of approximately 175,000 annual cases, a lower number than has been suggested in some other studies. Further preliminary analysis suggests there is a critical relationship between rapidity of antibiotic initiation and source control implementation following onset of hypotension and outcome in septic shock (Kumar et al, CCM 2006).

SECONDARY OUTCOMES:
Vasopressor use as a predictor of complications | Participants will be followed for the Average length of hospital stay 4-5 weeks
  1. utility of persistence or increase of vasopressor needs over the 1st 24 hours of shock as a predictor of a complicated ICU course (ICU duration > 1 week) or death.
  Captured in the data collection tool
Elements that predict complications in ICU | Participants will be followed for the Average length of hospital stay 4-5 weeks
  2.assessment of initial biochemical parameters, co-morbidities and new onset organ failure at admission as predictors of a complicated ICU course (ICU duration > 1 week) and death.
  Measured by the data collection tool

CONTACTS AND LOCATIONS:
Overall Officials: Anand Kumar, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Winnipeg, Manitoba, Canada